CLINICAL TRIAL: NCT01812473
Title: Impact of Hypoalbuminemia on Voriconazole Pharmacokinetics in Critically Ill Adult Patients.
Brief Title: Plasma Protein Binding Characteristics of Voriconazole
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML8949; 2013-000559-42 (EudraCT Number)
Record Dates: First submitted 2013-03-01; First posted 2013-03-18 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-03

CONDITIONS: Focus of the Study:Protein Binding Characteristics of Voriconazole.
Keywords: protein binding; voriconazole; pediatrics; hematology; intensive care; albumin; alpha-1-acid-glycoprotein
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum samples are obtained to determine the albumin and alpha-1-acid-glycoprotein level.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients admitted to the Intensive Care Unit: All patients admitted to the Intensive Care Unit, treated with voriconazole are eligible for the study.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — During the treatment of voriconazole, at steady plasma concentrations of voriconazole, one plasma sample and one serum sample are taken.

SUMMARY:
The purpose of this study is to investigate the influence of hypoalbuminemia on the protein binding characteristics of the antifungal drug voriconazole in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* treated with voriconazole

Exclusion Criteria:

* None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Vanstraelen, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Admitted to the ICU Not Treated With Voriconazole: Patients admitted to the intensive Care Unit, with varying levels of plasma albumin concentrations during admission.
  Plasma from this patients will be spiked in vitro with different voriconazole concentrations to investigate the influence of low albumine concentrations in plasma on voriconazole protein binding characteristics.
- Patients Admitted to the ICU Treated With Voriconazole: Patients admitted to the Intensive Care Unit, treated with voriconazole are included in this study. Voriconazole protein binding will be determined and the correlation with albumin plasma concentrations will be evaluated.
Period: Overall Study
Arm/Group | Patients Admitted to the ICU Not Treated With Voriconazole | Patients Admitted to the ICU Treated With Voriconazole
Started | 22 | 13
Completed | 22 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Admitted Tot the ICU Not Treated With Voriconazole: Patients admitted to the intensive Care Unit, with varying levels of plasma albumin concentrations during admission.
  Plasma from this patients will be spiked in vitro with different voriconazole concentrations to investigate the influence of low albumine concentrations in plasma on voriconazole protein binding characteristics.
- Total: Total of all reporting groups
Arm/Group | Patients Admitted Tot the ICU Not Treated With Voriconazole | Patients Admitted to the ICU Treated With Voriconazole | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 74] | 62 [57.5 to 71.5] | 65 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 14 | 7 | 21
Body weight [Median (Inter-Quartile Range); unit: kilogram] | 71 [60.3 to 80] | 68 [61 to 82.5] | 68 [62 to 80]
Acute Physiology and Chronic Health Evaluation (Apache) score [Mean (Standard Deviation); unit: units of the Apache Scoring system] — Calculated as the sum of all parameters described below. Every parameter is scored a value of 0 to +4, 0 being normal +4 being very high or low abnormal. The total apache score ranges from 0 to 71, with higher values being associated with more severe disease and higher mortality risk.
  Parameters included:Pa02 (arterial blood oxygen tension), rectal body temperature, Mean arterial pressure, arterial pH, heart rate, respiratory rate, serum sodium, serum potassium, serum creatinine, hematocrit, white blood cell count, glasgow coma scale.
  units of the Apache Scoring system | 23.5 (10) | 26.8 (6.9) | 25.3 (8.3)
Albumin plasma concentration [Median (Full Range); unit: gram/liter] | 23.7 [14.4 to 33.7] | 31.1 [13.8 to 38.7] | 26.7 [13.8 to 38.7]
alfa-1-acid glycoprotein plasma concentration [Median (Full Range); unit: gram/liter] | 1.4 [0 to 2.4] | 1.8 [1.1 to 3] | 1.5 [0 to 3.0]
Total plasma protein concentration [Mean (Standard Deviation); unit: gram/liter] | 53.4 (12.4) | 56.6 (7.3) | 54.2 (11.5)
Total plasma bilirubin concentration [Median (Inter-Quartile Range); unit: milligram/liter] | 0.75 [0.42 to 1.93] | 0.41 [0.28 to 1.69] | 0.67 [0.42 to 1.80]
Blood Urea Nitrogen [Median (Inter-Quartile Range); unit: milligram/deciliter] | 54.5 [37 to 146] | 70 [44.8 to 112.5] | 57.5 [37 to 132.5]
Creatinin plasma concentration [Median (Inter-Quartile Range); unit: milligram/deciliter] | 1.14 [0.67 to 1.99] | 0.95 [0.52 to 1.57] | 1.13 [0.67 to 1.81]
estimated Glomerular Filtration Rate (CKD-EPI equation) [Median (Inter-Quartile Range); unit: ml/min * 1.73m²] | 66 [40 to 93] | 84 [37.5 to 108.3] | 74 [40 to 100]
C reactive protein plasma concentration [Median (Inter-Quartile Range); unit: milligram/liter] | 72.1 [48.2 to 89.6] | 47.2 [21.6 to 116.9] | 71.5 [30.8 to 92.5]
Voriconazole daily dose [Median (Inter-Quartile Range); unit: milligram/kilogram/day] | NA [NA to NA] — Plasma from ICU patients was spiked with 1.5, 2.9 and 9 milligram/liter of voriconazole. | 8 [7.5 to 8.3] | NA [NA to NA] — In study A: Plasma from ICU patients was spiked with 1.5, 2.9 and 9 milligram/liter of voriconazole.
Total voriconazole plasma concentration [Median (Inter-Quartile Range); unit: milligram/liter] | NA [NA to NA] — Plasma was spiked with 1.5, 2.9 and 9 milligram/liter voriconazole | 2.4 [1.5 to 4.5] | 2.9 [1.5 to 9]
Unbound voriconazole plasma concentration [Median (Inter-Quartile Range); unit: milligram/liter] | 0.86 [0.45 to 2.66] | 0.71 [0.51 to 1.46] | 0.85 [0.46 to 2.55]
Bound voriconazole plasma concentration [Median (Inter-Quartile Range); unit: milligram / liter] | 1.63 [0.85 to 5.35] | 1.52 [1.07 to 2.57] | 1.62 [0.87 to 5.07]
Number of coadministered drugs bound to proteins for more then 70% [Mean (Inter-Quartile Range); unit: number of coadministered drugs] | 4.5 [1 to 6] | 2.5 [2 to 3] | 3 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Differences in Overall Protein Binding in the Presence of Different Plasma Albumin Concentrations.
Description: At steady state plasma concentrations of voriconazole, a plasma sample is taken to determine the overall protein binding of voriconazole. Equilibrium dialysis is used, followed by liquid chromatography-mass spectrometry.
Time Frame: At steady state plasma concentration of voriconazole (after day 4 of therapy)
Measure: Median (Inter-Quartile Range); unit: % of plasma protein binding
Units Other Than Participants: Plasma samples
Arm/Group | Patients Admitted Tot the ICU Not Treated With Voriconazole | Patients Admitted to the ICU Treated With Voriconazole
Number analyzed (Participants) | 22 | 13
Number analyzed (Plasma samples) | 66 | 20
% of plasma protein binding | 49.1 [42.6 to 52.3] | 49.6 [42.5 to 52.5]

ADVERSE EVENTS:
Arm/Group | Patients Admitted Tot the ICU Not Treated With Voriconazole | Patients Admitted to the ICU Treated With Voriconazole
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/13
Other Adverse Events (participants affected / at risk) | 0/22 | 0/13

LIMITATIONS AND CAVEATS:
Relatively small data set.

Only adult ICU patients.

No data are available for plasma albumin concentrations above 40 g/liter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No